CLINICAL TRIAL: NCT07109804
Title: Cuneiform Nucleus (CnF) Deep Brain Stimulation for Gait Facilitation Following Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Miami Project to Cure Paralysis (Other); Florida (Other)
Responsible Party: Principal Investigator, Brian Ronald Noga, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20240334; GR025072 (Other Grant/Funding Number: State of Florida)
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; deep brain stimulation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Deep Brain Stimulation (DBS) (Experimental): Participants will be in the DBS study group for up to 34 weeks.
  Interventions: Device: Deep Brain Stimulation (DBS); Procedure: Deep Brain Stimulation (DBS) Device Implant Procedure; Other: Training Sessions

INTERVENTIONS:
Device: Deep Brain Stimulation (DBS) — The DBS system delivers electrical current into deep areas of the brain. In this study, the electrical current will be delivered continuously during the study duration to an area of the brain called the cuneiform nucleus (CnF). Stimulation frequencies are anticipated to be between 20 and 50 Hertz. Participants may choose to continue stimulation following study termination. This area of the brain is associated with the body's ability to start a movement.
Procedure: Deep Brain Stimulation (DBS) Device Implant Procedure — Participants will undergo a one-time implantation of Cartesia DBS electrodes (bilateral) including the Vercise pulse generator in a single surgery (up to approximately 6 hours) to implant bilateral directional DBS leads in the cuneiform nucleus.
Other: Training Sessions — Training sessions occurs 3 times/week at the study center to condition the subjects before DBS implantation and after DBS implantation. Each session may last up to 60 minutes. Training sessions include joint mobility (passive stretching), volitional neuromuscular activation (active hip mobility), task isolation (weight shifting), task integration (stepping), and activity rehearsal (walking).

SUMMARY:
This is a study about deep brain stimulation (DBS) as an investigational treatment for walking impairment following spinal cord injury (SCI). The purpose of this study is to assess the feasibility and inform on the safety, and efficacy of CnF DBS to improve gait in SCI patients with incomplete injury who cannot effectively walk overground

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between ages of 22-70
* At least 1 year post SCI
* Confirmed SCI according to SCI clinician according to clinical history and the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) / American Spinal Injury Association (ASIA) criteria as documented in the American Spinal Injury Association Impairment Scale (AIS) on examination. Other disorders of gait will be excluded by history and a neurological examination.
* Persons with incomplete injury grades of ASIA C or D who can stand with support and who have some voluntary leg function and a maximum walking capacity of Walking Index for spinal cord injury - level II (WISCI-II) level 8 or less.
* Injury level T10 and above.
* Ability to stand with moderate body weight support for at least 5 minutes.
* Stable medical and physical condition.
* Able to commit to training/evaluation sessions over 6 months and for longer periodic follow-up.

Exclusion Criteria:

* Individuals with high-moderate to severe depression -Beck Depression Inventory II (BDI II) ≥ 25).
* Individuals with cognitive impairment indicated by a score of less than 24 on the Folstein Mini-Mental State Examination 2nd ed. (MMSE).
* Individuals with alcohol use disorder. The Alcohol Use Disorder Identification Test (AUDIT) will be used to measure harmful patterns of alcohol consumption over the past year. A cutoff score of 8 will be used to identify and exclude those with moderate to severe alcohol use behavior.
* Individuals with substance abuse. The Drug Abuse Screening Test (DAST-10) will be used to identify problematic substance abuse behavior over the past year. A cutoff score of 6 will be used to identify and exclude those with moderate to severe drug use behavior.
* The presence of major medical co-morbidities and other surgical contra-indications such as coagulopathy as defined by past medical history and abnormal lab work at the investigator/surgeon's discretion.
* Individuals with a Berg Balance score < 21.
* Individuals with a history of traumatic brain injury (TBI), seizures, severe autonomic dysreflexia, dysphagia or osteoporosis.
* History of prior intracranial surgery or known lesions.
* Individuals that require diathermy, repetitive transcranial magnetic stimulation, electroconvulsive therapy, or serial brain MRIs.
* Individuals with non-MRI compatible metallic implants in their head or body, and with metallic implants and other implantable devices in the body that could be affected by DBS.
* Individuals with active implantable devices anywhere in the body (e.g., cardiac pacemaker, defibrillator, implanted medication pump).
* Individuals who are pregnant desire to become pregnant during the study.
* Individuals who are breastfeeding.
* Individuals with intractable orthostatic hypotension despite treatment.
* Individuals with a recent history of limb fracture, ligamentous injury, active pressure sores or unstable skin structures (e.g., skin grafts and chest tubes).

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in walking speed measured by 10-meter walk test | baseline, up to 34 weeks
  The ten-meter walk test will be measured in meters/second.
Change in distance measured by 6-min walk test | baseline, up to 34 weeks
  The 6-min walk test will be measured in meters

CONTACTS AND LOCATIONS:
Overall Officials: Brian R Noga, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - The Miami Project to Cure Paralysis, Miami, Florida
  - University of Miami School Of Medicine, Miami, Florida

IPD SHARING:
Plan to Share IPD: No